CLINICAL TRIAL: NCT07208968
Title: Metal Artifact Reduction Sequence MRI for Surgical Decision-Making in Infected Unicompartmental Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Xinyu Fang, Deputy chief physician, First Affiliated Hospital of Fujian Medical University
Other Study IDs: MTCA,ECFAH Of FMU [2015]084 -1
Record Dates: First submitted 2025-09-21; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Prosthetic Joint Infection; Unicompartmental Knee Arthroplasty
Keywords: Prosthetic joint infection; Unicompartmental knee arthroplasty; Antibiotics and implant retention; One-stage revision; Unicompartmental spacer; Metal artefact reduction sequence magnetic resonance imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DAIR group: Patients with acute/hematogenous uPJI underwent debridement, antibiotics and implant retention (DAIR)
- Revision group: Patients with chronic uPJI underwent revision.

SUMMARY:
A single-center retrospective cohort study was conducted in the Department of Orthopedics of Fujian Medical University Affiliated First Hospital. This study reviewed 28 patients who received unicompartmental prosthetic joint infection (uPJI) treatment at this institution from 2017 to 2023. The personal information of the patients, including age, gender, affected side, age-adjusted Charles Syndrome Index (aCCI), inflammation markers, lesion range on magnetic resonance angiography (MARS-MRI), lesion range observed directly during surgery and surgical methods, were recorded in detail. The study evaluated the clinical decision-making of a standardized MARS-MRI-guided treatment protocol for uPJI by reviewing the clinical outcomes of uPJI patients in a single PJI center.

DETAILED DESCRIPTION:
A single-center retrospective cohort study was conducted in the Department of Orthopedics of Fujian Medical University Affiliated First Hospital. This study reviewed 28 patients who received unicompartmental prosthetic joint infection (uPJI) treatment at this institution from 2017 to 2023. The personal information of the patients, including age, gender, affected side, age-adjusted Charles Syndrome Index (aCCI), inflammation markers, lesion range on magnetic resonance angiography (MARS-MRI), lesion range observed directly during surgery and surgical methods, were recorded in detail. The study evaluated the clinical decision-making of a standardized MARS-MRI-guided treatment protocol for uPJI by reviewing the clinical outcomes (infection control and functional recovery) of uPJI patients in a single PJI center.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of uPJI on the basis of medical history, symptoms, imaging data, etc.;
2. Treatment by internal fixation surgery;
3. Normal cognitive function;
4. Informed consent obtained from the patient or family.

Exclusion Criteria:

1. Significant missing data: In accordance with the Transparent Reporting of a Multivariate Prediction Model for Individual Prognosis or Diagnosis (TRIPOD) statement, only cases with complete key variables (missing rate <5%) were included;
2. Severe preoperative systemic comorbidities (e.g., decompensated liver/renal failure, active pneumonia, malignancy, and cachexia) and/or a history of mental illness;
3. Missing postoperative follow-up.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty-seven patients (28 knees) diagnosed with uPJI from 2017 to 2024 were analyzed. MARS-MRI and intraoperative direct vision were used to confirm the extent of lesions. All patients completed at least one year of follow-up. Follow-up comprised comprehensive orthopaedic examinations and serological tests, supplemented by repeat imaging where necessary to assess local fracture/internal fixation status.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Infection control or not according to the MSIS criteria | preoperative and two-year follow-up
  According to the Musculoskeletal Infection Society (MSIS) criteria, infection control was defined as no local inflammation, infection/aseptic revision, or uPJI-related death within 1 year of the initial surgery.
The Hospital for Special Surgery Knee Score (HSS) score | preoperative and two-year follow-up
  The Hospital for Special Surgery Knee Score (HSS) is a patient-reported questionnaire specific to the knee joint, with a total score of 100 points. It comprises six scoring components: pain (30 points), function (22 points), range of motion (18 points), muscle strength (10 points), knee deformity (10 points) and stability (10 points). Additional points are deducted for the use of assistive devices, extension lag and varus deformity: up to 3 points for assistive device use, up to 5 points for extension lag and 1 point deducted for every 5 degrees of varus deformity. The scores are classified as follows: ≥ 85 as "Excellent", 70-84 as "Good", 60-69 as "Fair", and < 60 as "Poor". The HSS score is widely praised for its perceived ease of use and quick recording and has been shown to be an effective and reliable measure for assessing the efficacy of TKA.

SECONDARY OUTCOMES:
Range of motion | preoperative and two-year follow-up
Visual Analogue Scale (VAS) score | preoperative and two-year follow-up
  VAS scores are the most commonly used indicator for assessing the intensity of patient pain. The scale ranges from "0" to "10", where "0" indicates no pain and "10" represents the most severe pain that is unbearable. Patients will rate their pain based on subjective perceptions. In this trial, VAS scores will be recorded once before TKA. The VAS scores will be assessed separately for the resting and flexion states. If the patient's hospitalization period is shorter than 72 hours, the VAS score at discharge will be recorded instead of that at 72 hours. Studies have shown that some patients still experience joint pain six months after TKA. The VAS scores of patients at 6 months after TKA will be evaluated. A VAS score of 4 or above is defined as "chronic persistent pain after TKA." The results will be used to evaluate whether PSIA can reduce pain after TKA.
Pathogens Type | preoperative and two-year follow-up
  The pathogen that caused the patient's current infection was finally identified through culture.
SF-12 score | preoperative and two-year follow-up
  SF-12 (12-Item Short Form Health Survey) is a health-related quality of life (HRQoL) assessment tool. It consists of 12 items, mainly covering two core aspects: PCS (Physical Component Summary, summary of physical health) and MCS (Mental Component Summary, summary of mental health). The dimensions covered include: physical function (PF), limitations in daily activities (RP), physical pain (BP), overall health (GH), vitality (VT), social function (SF), emotional role function (RE), and mental health (MH). It enables the assessment of patients' overall health status within a relatively short period of time. It is often used to evaluate the changes in patients' quality of life before and after orthopedic surgeries (such as joint replacement, spinal surgery, ligament reconstruction, etc.). The range value is 0 to 100. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China